CLINICAL TRIAL: NCT00984009
Title: A One-Directional, Open-Label Drug-Food Interaction Study to Investigate the Effects of Multiple-Daily Consumptions of Grapefruit Juice on the Single-Dose Pharmacokinetics of Colchicine in Healthy Volunteers
Brief Title: A Drug-Food Interaction Study Between Colchicine and Grapefruit Juice
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-08-1017
Record Dates: First submitted 2009-08-13; First posted 2009-09-24 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Pharmacokinetics
Keywords: healthy; pharmacokinetics; grapefruit juice; furanocoumarins; cytochrome p450 3A4
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine alone (Active Comparator): baseline colchicine pharmacokinetics
  Interventions: Drug: Colchicine
- Colchicine with Grapefruit Juice (Experimental): colchicine pharmacokinetics in presence of grapefruit juice
  Interventions: Other: Grapefruit Juice; Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — A single dose of 0.6 mg colchicine administered alone at 7:15 a.m. on Day 1
  Other Names: COLCRYS™
  Arms: Colchicine alone
Other: Grapefruit Juice — 240 mL of grapefruit juice ingested twice daily at 7:15 a.m. and 7:15 p.m. on Days 15 to 18.
  Arms: Colchicine with Grapefruit Juice
Drug: Colchicine — A single dose of 0.6 mg colchicine administered with grapefruit juice at 7:15 a.m. on Day 18 after an overnight fast of at least 10 hours.
  Arms: Colchicine with Grapefruit Juice

SUMMARY:
Grapefruit juice is an inhibitor of the cytochrome P450 (CYP) 3A4 enzyme system, one of the enzyme systems responsible for the metabolism of colchicine. This study will evaluate the effect of multiple daily consumptions of grapefruit juice on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period.

DETAILED DESCRIPTION:
Grapefruit juice is an inhibitor of the cytochrome P450 (CYP) 3A4 enzyme system, one of the enzyme systems responsible for the metabolism of colchicine. This study will evaluate the effect of multiple daily consumptions of grapefruit juice on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. On study Day 1, after a fast of at least 10 hours twenty-two healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one dose of colchicine (1 x 0.6 mg tablet). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of colchicine. Blood sampling will continue on a non-confined basis on Days 2-5. After a 14 day washout period, starting on the morning of Day 15 and continuing through Day 17, subjects will return to the clinic for consumption of an administered dose of grapefruit juice (1 x 240 ml) twice daily. On the morning of Day 18 after a fast of at least 10 hours all subjects will receive a co-administered single oral dose of colchicine (1 x 0.6 mg) and grapefruit juice (1 x 240 ml). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of colchicine in the presence of grapefruit juice. Blood sampling will continue on a non-confined basis on Days 19-22. Subjects will consume the final administered dose of grapefruit juice (1 x 240 ml) in the evening on Day 18. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Seated blood pressure and pulse will be measured prior to dosing and at approximately 1, 2, and 3 hours following drug administration on Days 1 and 18 to coincide with peak plasma concentrations of colchicine. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age, non-smoking and non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures) with a body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive.

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to colchicine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm.D., Principal Investigator — PRACS - Cetero
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Wason S, DiGiacinto JL, Davis MW. Effects of grapefruit and Seville orange juices on the pharmacokinetic properties of colchicine in healthy subjects. Clin Ther. 2012 Oct;34(10):2161-73. doi: 10.1016/j.clinthera.2012.08.007. Epub 2012 Aug 31. PMID 22940371
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-two (22) healthy, non-smoking, non-obese, adult, male and female volunteers, consisting of members of the community at large, were enrolled in the study.
Pre-assignment Details: 46 subjects screened, 13 were screen failures, 6 had schedule conflicts or were no shows for check-in, 1 was not screened per request of study site, 2 were transferred to a different study
Groups:
- Colchicine Alone / With Grapefruit Juice: [All subjects received each of the study treatments.] Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:15 a.m. after an overnight fast, followed by a washout period of 14 days. On Days 15 to 17, each subject received one 240 ml serving of grapefruit juice twice daily, at 7:15 a.m. and 7:15 p.m, without regard to meals. Then, on Day 18, each subject received both one 0.6 mg colchicine tablet and one 240 ml serving of grapefruit juice at 7:15 a.m. after an overnight fast. A final 240 ml serving of grapefruit juice was administered at 7:15 p.m. that evening.
Period: Colchicine Alone
Arm/Group | Colchicine Alone / With Grapefruit Juice
Started | 22
Completed | 22
Not Completed | 0
Period: 14 Day Washout Period
Arm/Group | Colchicine Alone / With Grapefruit Juice
Started | 22
Completed | 22
Not Completed | 0
Period: Grapefruit Juice Alone
Arm/Group | Colchicine Alone / With Grapefruit Juice
Started | 22
Completed | 21 (one subject dropped due to missed a.m. serving of grapefruit juice on Day 16)
Not Completed | 1
Not completed — missed serving of grapefruit juice | 1
Period: Colchicine With Grapefruit Juice
Arm/Group | Colchicine Alone / With Grapefruit Juice
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colchicine Alone / With Grapefruit Juice
Number analyzed (Participants) | 22
Age, Customized [Number; unit: participants] — age range: ≥18 and ≤45
  participants
    <=18 years | 0
    Between 18 and 65 years | 22
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn immediately prior to colchicine dosing on Days 1 and 18, and then 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, and 96 hours after colchicine dose administration
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine Alone: Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:15 a.m. after an overnight fast, followed by a washout period of 14 days.
- Colchicine With Grapefruit Juice: On Days 15 to 17, each subject received one 240 ml serving of grapefruit juice twice daily, at 7:15 a.m. and 7:15 p.m, without regard to meals. Then, on Day 18, each subject received both one 0.6 mg colchicine tablet and one 240 ml serving of grapefruit juice at 7:15 a.m. after an overnight fast. A final 240 ml serving of grapefruit juice was administered at 7:15 p.m. that evening.
Arm/Group | Colchicine Alone | Colchicine With Grapefruit Juice
Number analyzed (Participants) | 21 | 21
pg/mL | 2,172.96 (652.99) | 1,971.10 (398.80)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable colchicine concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Grapefruit Juice
Number analyzed (Participants) | 21 | 21
pg-hr/mL | 9,329.53 (3,367.85) | 8,823.40 (3,003.15)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable colchicine plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Grapefruit Juice
Number analyzed (Participants) | 21 | 21
pg-hr/mL | 11,079.98 (3,949.27) | 10,854.22 (4,140.12)

ADVERSE EVENTS:
Groups:
- Grapefruit Juice Alone: On Days 15 to 17, each subject received one 240 ml serving of grapefruit juice twice daily, at 7:15 a.m. and 7:15 p.m, without regard to meals.
- Colchicine With Grapefruit Juice: On Day 18, each subject received both one 0.6 mg colchicine tablet and one 240 ml serving of grapefruit juice at 7:15 a.m. after an overnight fast. A final 240 ml serving of grapefruit juice was administered at 7:15 p.m. that evening.
Arm/Group | Colchicine Alone | Grapefruit Juice Alone | Colchicine With Grapefruit Juice
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 1 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Colchicine Alone | Grapefruit Juice Alone | Colchicine With Grapefruit Juice
diarrhea (Gastrointestinal disorders) | 0/22 (0) | 0/22 (0) | 1/21 (1)
headache (Nervous system disorders) | 1/22 (1) | 0/22 (0) | 0/21 (0)
cough (Nervous system disorders) | 0/22 (0) | 0/22 (0) | 1/21 (1)
chest congestion (Respiratory, thoracic and mediastinal disorders) | 0/22 (0) | 0/22 (0) | 1/21 (1)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/22 (0) | 0/22 (0) | 1/21 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days